CLINICAL TRIAL: NCT05968456
Title: Complexity and Frailty in Cardiothoracic and Vascular Anesthesia (CAfCA). Prospective Multicentric Observational Study
Acronym: CAfCA
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Responsible Party: Principal Investigator, Federico Piccioni, Head of Anesthesia Section 1, Istituto Clinico Humanitas
Other Study IDs: CAfCA-3366
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Frailty; Anesthesia; Thoracic Surgery; Cardiothoracic Surgery; Vascular Surgery; Comorbidities and Coexisting Conditions
Keywords: Frailty; Thoracic surgery; Cardiac Surgery; Vascular Surgery
MeSH Terms: conditions — Frailty | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Thoracic surgery: Patient undergoing thoracic surgery
  Interventions: Other: Data collection
- Cardiac surgery: Patient undergoing cardiac surgery
  Interventions: Other: Data collection
- Vascular surgery: Patient undergoing vascular surgery
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Observational study in patients undergoing thoracic, cardiac and vascular surgery.

SUMMARY:
Frailty is a multidimensional syndrome characterized by a decline in physiological homeostatic reserve, which translates into an increased susceptibility to adverse events and unfavorable outcomes following even small exposures to physical, physiological or psychosocial stress.

In the European population up to 69 years, the prevalence is generally 6,5%, beyond 85 years of age it exceeds 50% and reaches 65% in the over-ninety population. The prevalence of frailty in the surgical population varies, depending on the studies, from 10 to 40%. Frailty and its severity grade represent themselves noticeably as strong predictors of adverse postoperative outcomes. The strongest evidence of association is recorded between frailty and mortality at 30 days.

The purpose of this study is to describe the characteristics of patients undergoing anesthesia for cardiothoracic and vascular surgery, with a specific focus on frailty elements and associated comorbidities that necessitate surgery.

This data analysis will provide valuable insights into the interaction between frailty, multimorbidity, and the perioperative pathway of patients undergoing cardiothoracic and vascular anesthesia.

DETAILED DESCRIPTION:
The Western population is going through a rapid process of aging, which is of major relevance for perioperative medicine because it is associated with an increase of approximately 2,5 times in postoperative morbidity and mortality. Despite the clear association between advanced age and adverse outcomes, there is a significant variability of outcomes in older patients which is not explainable solely based on the differences in age and comorbidities. In this regard, frailty seems to play a key role to explain such variability. Frailty is a multidimensional syndrome characterized by a decline in physiological homeostatic reserve, which translates into an increased susceptibility to adverse events and unfavorable outcomes following even small exposures to physical, physiological or psychosocial stress. However, frailty has not to be considered exclusively in a geriatric context. Several studies conducted in intensive care and perioperative settings have observed a not negligible prevalence of frailty also in age groups below 65 years.

In the European population up to 69 years, the prevalence is generally 6,5%, beyond 85 years of age it exceeds 50% and reaches 65% in the over-ninety population. The prevalence of frailty in the surgical population varies, depending on the studies, from 10 to 40%. Such variability is determined by several factors: the tools and thresholds used to define frailty, the type of surgery, the type of procedure within the same surgical specialty and the setting of surgery. In cardiac surgery, prevalences oscillating between 10 and 50% have been reported. In vascular surgery, the prevalence of frailty is on average high oscillating between 20 and 60%, while in the field of thoracic surgery data of prevalence stands around 12 and 50%.

Frailty and its severity grade represent themselves noticeably as strong predictors of adverse postoperative outcomes. The strongest evidence of association is recorded between frailty and mortality at 30 days (Odds Ration variable between 1.4 and 8.33).

In the physio-pathological processes that link frailty to adverse postoperative outcomes, there are certainly modifiable factors. Several data in the literature demonstrate this correlation, including the evidence that patients diagnosed with frailty, if subjected to major elective surgery in centers with low volumes of fragile patients, have lower rates of survival at 30 days and a higher incidence of mortality correlated to postoperative complications, other conditions being equal.

From what has been outlined, it is easy to understand how a better knowledge of frailty and its prevalence can be useful for health systems that have to be more and more structured with the availability of clinical and organizational resources appropriate for the increasing complexity and frailty of patients.

The purpose of this study is to describe the characteristics of patients undergoing anesthesia for cardiothoracic and vascular surgery, with a specific focus on frailty elements and associated comorbidities that necessitate surgery.

This data analysis will provide valuable insights into the interaction between frailty, multimorbidity, and the perioperative pathway of patients. Additionally, it will facilitate the development of a comprehensive description of clinical and organizational resources and their utilization in managing this specific category of patients.

This study will lay the foundations for further, more specific studies in this field and will provide useful information to build more suitable anesthesiologic clinical care pathways for the increasing demands of fragile and complex patients.

STUDY DESIGN

The study will be prospective, multicentric observational at the national level.

Data collection will not modify anesthetic treatments for patients included in the study or their treatment pathways. Therefore, according to current legislation, a conclusion of ad hoc insurance policies is not necessary.

Anthropometric, functional and procedural data will be collected during the pre-, intra- and post-operative period.

The period of observation for each enrolled subject starts with the first pre-operative anesthesiology assessment and ends 30 days after surgical intervention. Data relative to preoperative condition, surgical preparation and intra- and post-operative information of the subject will be collected.

Data collection will be constituted by a common part including all patients (CAfCA core) and specific parts related to the fields of cardiac, thoracic and vascular surgery aimed to specifically characterize these subgroups of patients.

SAMPLE SIZE

This research is a prospective pilot study aiming at studying patients subjected to cardiac-thoracic-vascular surgery. In this field, very heterogeneous data has been reported in terms of frailty prevalence, as mentioned in the introduction, which varies between 20% and 60% according to which study is considered.

Considering a conservative estimation of the frailty prevalence of 50%, a margin of error and a population of 380 patients is sufficient to estimate the prevalence of frailty in the cardiac-thoracic-vascular population with a 95% confidence interval. This number is increased by 5% for a total of 400 patients to take account of missing data and drop-out. To reliably estimate the prevalence of frailty not only in the general cardiac-thoracic-vascular population, but also - as the secondary outcome - in each of the 3 subpopulations, meaning the prevalence of frailty in cardiac, thoracic and vascular surgery, a sample of 500 patients will allow answering both to the primary outcome of frailty prevalence in the general population and to the secondary outcome of prevalence in the 3 subpopulations. For this purpose, it is supposed that every subgroup will contribute with 1/3 of the total enrolled patients (i.e. 166 patients) and, keeping a conservative estimate of the prevalence of 50%, in this case, the sample is sufficient to estimate frailty prevalence with a 7.5% margin of error in each of the 3 subpopulations, with a confidence interval of 95%.

Considering the observational nature of the study, the protocol allows for the possibility of recruiting a larger number of patients if the participating centers are willing to do so. By increasing the sample size, the study can achieve a higher level of precision in estimating the prevalence of frailty within the investigated subpopulations.

CLINICAL MANAGEMENT

During the preoperative anesthesiologic assessment, every eligible patient will be provided with a detailed explanation of the study protocol. They will be given the opportunity to review the study information and, if willing to participate, a signed informed consent will be obtained. Enrollment can take place during the pre-operative assessment or after the patient's admission to the hospital.

It is important to note that participating patients have the right to withdraw from the study at any time.

During enrolment, patients will be subjected to tests evaluating pharmacologic therapy adherence (Morinsky scale - MMAS-8), frailty evaluation test (Clinical Frailty Scale - CFS, Tilburg Frailty Indicator - TFI, Modified Frailty Index both the 5 and 11 items versions - mFI-5 and mFI-11) and engagement evaluation tests (Patient Health Engagement - PHE score).

Furthermore, for each patient, the ASA score, Charlson comorbidity score, MUST score, ACS NSQIP, physiologic P-POSSUM, Revised Cardiac Risk Index (RCRI), AKI risk index and ARISCAT score will be registered.

Other evaluation scores will be employed specifically for the different patient types:

* Cardiac surgery patients: EUROSCORE II and FORECST (evaluation of frailty in cardiac surgery)
* Thoracic surgery patients: ThRCRI, Thoracoscore, Eurolung 1 and 2, ECOG performance status scale
* Vascular surgery patients: V-Possum

The data retrieved through the aforementioned scores will not be utilized to modify the patients' perioperative pathway unless they are already part of specific protocols implemented by the participating center. The surgical and anesthesiologic procedures will be conducted according to the local management protocols, and participation in the study will not result in any modifications to these procedures.

The experimenters at each center will be limited to reporting the patients' preoperative clinical conditions, laboratory and instrumental exams, information regarding the performed surgery, and any complications that occur during the hospital stay.

The experimenter will conduct re-evaluations of each patient from the first to the fifth postoperative day, as well as at the time of hospital discharge, in order to record any potential medical or surgical complications that may arise. Additionally, a follow-up will be conducted 30 days after discharge via phone to assess the patient's health status and record any incidences of complications, re-hospitalization, or mortality.

Complications will be recorded in a specific manner, utilizing the Clavien-Dindo classification system. This classification system provides standardized criteria for defining and grading complications. The definitions of complications will be based on established guidelines and international consensus documents published in the literature, ensuring consistency and accuracy in the recording and reporting of complications throughout the study.

DATA GATHERING AND ANALYSIS PLAN

Data will be retrieved in pseudo-anonym form. Data gathering will be made through a specifically created database, on RedCap platform, which has been made available by the Italian Society of Anesthesiology and Intensive Care Medicine (Società Italiana di Anestesia Analgesia Rianimazione e Terapia Intensiva - SIAARTI).

Analysis Plan No interim analyses are expected. Most of the statistical analysis will be descriptive. Categorical variables considered will be described in terms of frequency and percentages, and continuous variables in terms of mean (sd) and median (IQR) as appropriate. The primary objective will be described in terms of prevalence with 95% of the expected confidence interval.

Univariate comparative analyses will be conducted through Chi-Square test and Mann-Whitney U-test as appropriate, considering a significance level of 0.05 in the general population and stratifying the 3 populations. Missing data will be analyzed and handled if necessary, with multiple-imputation or analog techniques.

The correlation between frailty scores will be investigated through Bland-Altman analysis and correlation coefficient.

A multivariate correlation analysis will be conducted to explore associations between preoperative factors, pre-operative risk scores, frailty and outcomes.

The possibility to perform further analyses non specified in the protocol but suggested by the above-mentioned planned analyses is admitted (particularly in the cardiac-thoracic-vascular filed of the three subgroups of patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiac, thoracic or vascular surgery
* Patients aged 18 or older
* Patients who have provided informed consent to participate in the study.

Exclusion Criteria:

* Patients subjected to surgery in urgency and emergency settings
* Procedures in one-day surgery settings
* Procedures without the involvement of anesthesiologists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to anesthesia for elective cardiac-thoracic-vascular surgery consecutively recruited during a period of 1 month designated by each partecipating center
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Frailty Prevalence | at preoperative evaluation visit
  Determine the prevalence of frailty in the sample using the Clinical Frailty Score, in the three clinical areas: cardiac, thoracic, and vascular surgery
Frailty Prevalence comparison | at preoperative evaluation visit
  Frailty prevalence comparison among the three clinical areas: cardiac, thoracic, and vascular surgery

SECONDARY OUTCOMES:
Frailty assessment instruments comparison | at preoperative evaluation visit
  Agreement between different frailty instruments
Multimorbidity description | at preoperative evaluation visit
  Describe the multimorbidity profile of the included patients.
In-hospital complications | up to 30 days after operation
  Incidence of in-hospital complications
Unplanned ICU admission | up to 30 days after operation
  Unplanned ICU admissions rate
Length of hospital stay | up to 30 days after operation
  Length of hospital stay (days)
In-hospital mortality | up to 30 days after operation
  In-hospital mortality rate
30-day mortality | up to 30 days after operation
  Mortality rate at 30 days after intervention
Association between different frailty risk scores and clinical outcomes | up to 30 days after operation
  Association between different frailty risk scores and clinical outcomes (complications, length of stay, mortality)
Correlation between perioperative risk scores and frailty scores | at preoperative evaluation visit
  Correlation between perioperative risk scores and frailty scores
Description of the perioperative clinical pathway | up to 30 days after operation
  Describe the perioperative clinical care pathway followed by the enrolled subjects
Description of the anesthesiologic techniques adopted | up to 30 days after operation
  Provide details on the anesthesiologic techniques utilized and the level of invasiveness of hemodynamic monitoring employed.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Piccioni, Dr, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (8):
- Italy (8):
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Spedali Civili di Brescia, Brescia
  - ASST Ovest Milanese, Legnano
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - AOR San Carlo, Potenza
  - Azienda Ospedaliero Universitaria Senese, Siena
  - Azienda Ospedaliera Umberto I Mauriziano, Turin
  - Città della salute e della Scienza di Torino, Turin

REFERENCES:
- [Background] Fowler AJ, Abbott TEF, Prowle J, Pearse RM. Age of patients undergoing surgery. Br J Surg. 2019 Jul;106(8):1012-1018. doi: 10.1002/bjs.11148. Epub 2019 May 22. PMID 31115918
- [Background] Hamel MB, Henderson WG, Khuri SF, Daley J. Surgical outcomes for patients aged 80 and older: morbidity and mortality from major noncardiac surgery. J Am Geriatr Soc. 2005 Mar;53(3):424-9. doi: 10.1111/j.1532-5415.2005.53159.x. PMID 15743284
- [Background] Turrentine FE, Wang H, Simpson VB, Jones RS. Surgical risk factors, morbidity, and mortality in elderly patients. J Am Coll Surg. 2006 Dec;203(6):865-77. doi: 10.1016/j.jamcollsurg.2006.08.026. PMID 17116555
- [Background] Oresanya LB, Lyons WL, Finlayson E. Preoperative assessment of the older patient: a narrative review. JAMA. 2014 May;311(20):2110-20. doi: 10.1001/jama.2014.4573. PMID 24867014
- [Background] McIsaac DI, MacDonald DB, Aucoin SD. Frailty for Perioperative Clinicians: A Narrative Review. Anesth Analg. 2020 Jun;130(6):1450-1460. doi: 10.1213/ANE.0000000000004602. PMID 32384334
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Koh LY, Hwang NC. Frailty in Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):521-531. doi: 10.1053/j.jvca.2018.02.032. Epub 2018 Feb 22. No abstract available. PMID 29580797
- [Background] Gale CR, Cooper C, Sayer AA. Prevalence of frailty and disability: findings from the English Longitudinal Study of Ageing. Age Ageing. 2015 Jan;44(1):162-5. doi: 10.1093/ageing/afu148. Epub 2014 Oct 12. PMID 25313241
- [Background] McIsaac DI, Wijeysundera DN, Huang A, Bryson GL, van Walraven C. Association of the Hospital Volume of Frail Surgical Patients Cared for with Outcomes after Elective, Major Noncardiac Surgery: A Retrospective Population-based Cohort Study. Anesthesiology. 2017 Apr;126(4):602-613. doi: 10.1097/ALN.0000000000001536. PMID 28157134
- [Background] Lee JA, Yanagawa B, An KR, Arora RC, Verma S, Friedrich JO; Canadian Cardiovascular Surgery Meta-Analysis Working Group. Frailty and pre-frailty in cardiac surgery: a systematic review and meta-analysis of 66,448 patients. J Cardiothorac Surg. 2021 Jun 25;16(1):184. doi: 10.1186/s13019-021-01541-8. PMID 34172059
- [Background] Sivaharan A, Boylan L, Witham MD, Nandhra S; Northern Vascular Centre. Sarcopenia in Patients Undergoing Lower Limb Bypass Surgery is Associated with Higher Mortality and Major Amputation Rates. Ann Vasc Surg. 2021 Aug;75:227-236. doi: 10.1016/j.avsg.2021.02.022. Epub 2021 Apr 2. PMID 33819585
- [Background] Tsiouris A, Hammoud ZT, Velanovich V, Hodari A, Borgi J, Rubinfeld I. A modified frailty index to assess morbidity and mortality after lobectomy. J Surg Res. 2013 Jul;183(1):40-6. doi: 10.1016/j.jss.2012.11.059. Epub 2012 Dec 21. PMID 23273884
- [Background] Beckert AK, Huisingh-Scheetz M, Thompson K, Celauro AD, Williams J, Pachwicewicz P, Ferguson MK. Screening for Frailty in Thoracic Surgical Patients. Ann Thorac Surg. 2017 Mar;103(3):956-961. doi: 10.1016/j.athoracsur.2016.08.078. Epub 2016 Oct 6. PMID 27720368
- [Background] Handforth C, Clegg A, Young C, Simpkins S, Seymour MT, Selby PJ, Young J. The prevalence and outcomes of frailty in older cancer patients: a systematic review. Ann Oncol. 2015 Jun;26(6):1091-1101. doi: 10.1093/annonc/mdu540. Epub 2014 Nov 17. PMID 25403592
- [Background] Lin HS, Watts JN, Peel NM, Hubbard RE. Frailty and post-operative outcomes in older surgical patients: a systematic review. BMC Geriatr. 2016 Aug 31;16(1):157. doi: 10.1186/s12877-016-0329-8. PMID 27580947
- [Background] Stortecky S, Schoenenberger AW, Moser A, Kalesan B, Juni P, Carrel T, Bischoff S, Schoenenberger CM, Stuck AE, Windecker S, Wenaweser P. Evaluation of multidimensional geriatric assessment as a predictor of mortality and cardiovascular events after transcatheter aortic valve implantation. JACC Cardiovasc Interv. 2012 May;5(5):489-496. doi: 10.1016/j.jcin.2012.02.012. PMID 22625186
- [Background] Velanovich V, Antoine H, Swartz A, Peters D, Rubinfeld I. Accumulating deficits model of frailty and postoperative mortality and morbidity: its application to a national database. J Surg Res. 2013 Jul;183(1):104-10. doi: 10.1016/j.jss.2013.01.021. Epub 2013 Feb 1. PMID 23415494